CLINICAL TRIAL: NCT06460831
Title: A Comparative Study Evaluating the Vein of MArshall Ethanol Infusion Ablation Using an Over-the-wire (OTW) Balloon Versus a microcatHeter in Patients With Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Chief of the Arrhythmia Center, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MARSHALL-CATH study
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: marshall vein; mitral valve isthmus line
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OTW group (Placebo Comparator)
  Interventions: Device: OTW
- Microcatheter group (Experimental)
  Interventions: Device: Microcatheter

INTERVENTIONS:
Device: Microcatheter — The microcatheter group undergoes alcohol ablation using a microcatheter.
  Arms: Microcatheter group
Device: OTW — The OTW group undergoes alcohol ablation using an OTW balloon.
  Arms: OTW group

SUMMARY:
The goal of this study is to compare OTW balloon with microcatheter in the Marshall vein alcohol ablation study. The main questions it aims to answer are: • Is there a difference in the effectiveness and safety of OTW balloon and microcatheter in Marshall vein alcohol ablation? Participants will be asked to:

Undergo treatment with OTW balloon Undergo treatment with microcatheter If there is a comparison group: Researchers will compare the OTW balloon group and the microcatheter group to see different effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-80 years.
2. Persistent atrial fibrillation or atrial flutter dependent on the mitral isthmus.
3. Inadequate response to antiarrhythmic drug therapy, or intolerance to antiarrhythmic drugs.
4. New York Heart Association functional class ≤ IV,with left ventricular ejection fraction (LVEF) ≥ 35%

Exclusion Criteria:

1. Patients with known allergies to alcohol.
2. Participants with a history of serious cardiovascular events such as myocardial infarction or stroke within the past three months will be excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute rate of mitral isthmus block | During catheter ablation procedures
  Efficacy endpoints
Procedural complications | During catheter ablation procedures
  Safety endpoints
Recovery rate of the mitral isthmus line | beyond 3 months after the ablation procedure.
  Long-term primary efficacy endpoints

SECONDARY OUTCOMES:
Procedural characteristics | Periprocedural period
Hospitalization costs | Periprocedural period

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Ren Ji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Yuhuan Second People's Hospital, Taizhou, Zhejiang
  - Changshu Hospital of Traditional Chinese Medical, Changshu

IPD SHARING:
Plan to Share IPD: Undecided